CLINICAL TRIAL: NCT03760796
Title: The Johns Hopkins Myocardial Infarction, COmbined-device, Recovery Enhancement (MiCORE) Study
Brief Title: Myocardial Infarction, COmbined-device, Recovery Enhancement Study
Acronym: MiCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Apple Inc. (Industry); iHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00099938
Record Dates: First submitted 2018-11-21; First posted 2018-11-30 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction
Keywords: readmission; cardiovascular disease prevention; cardiovascular disease risk factors; cost-effectiveness; heart attack; acute myocardial infarction; secondary prevention; digital health; smartphone app; self-management; guideline adherence; behavior modification
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Single group assignment to the Corrie Health Digital Platform prospective intervention group (n=200), as compared with a historical standard of care comparison group (n=864)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Corrie Health Digital Platform group (Experimental): Receives the Corrie Health intervention plus the standard of care
  Interventions: Device: Corrie Health Digital Platform

INTERVENTIONS:
Device: Corrie Health Digital Platform — The Corrie Health Digital Platform consists of the Corrie smartphone app for heart attack recovery which is paired with an Apple Watch and Bluetooth-enabled, iHealth blood pressure monitor.

SUMMARY:
Unplanned readmissions after hospitalization for acute myocardial infarction (AMI) are among the leading causes of preventable morbidity, mortality, and healthcare costs. Digital health interventions (DHI) could be an effective tool in promoting self-management, adherence to guideline directed therapy, and cardiovascular risk reduction.

A DHI developed at Johns Hopkins-the Corrie Health Digital Platform-includes the first cardiology Apple CareKit smartphone application, paired with an Apple Watch and iHealth Bluetooth-enabled blood pressure monitor. Corrie targets: (1) self-management of cardiac medications, (2) self-tracking of vital signs, (3) education about cardiovascular disease through articles and animated videos, and (4) care coordination that includes cardiac rehabilitation and outpatient follow-up appointments.

In this prospective study, STEMI or type 1 NSTEMI patients are being enrolled to use the Corrie Health Digital Platform beginning early during participants' hospital stay. Enrollment sites include Johns Hopkins Hospital, Johns Hopkins Bayview Medical Center, Massachusetts General Hospital, and Reading Hospital. The primary objective is to compare time to first readmission within 30 days post-discharge among patients with the Corrie Health Digital Platform to patients in the historical standard of care comparison group.

ELIGIBILITY:
Corrie Health Digital Platform group

Inclusion Criteria:

* Admitted for acute myocardial infarction (STEMI or Type 1 NSTEMI)
* 18 years or older
* English-speaking
* Own any type of smartphone

Exclusion Criteria:

* Visual, hearing, or motor impairment which precludes the use of the intervention
* Inability to participate due to severity of illness (e.g., intubated and on sedation in the setting of cardiogenic shock). If patients are deemed clinically unstable and unable to participate at the time of initial screening, the research team member returns at a later date to determine whether this status has changed.

Historical Standard of Care Comparison group

Inclusion Criteria:

* Admitted for acute myocardial infarction (STEMI or NSTEMI)
* 18 years or older
* English-speaking

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth S Martin, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Reading Hospital-Tower Health, Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaulding EM, Marvel FA, Lee MA, Yang WE, Demo R, Wang J, Xun H, Shah L, Weng D, Fashanu OE, Carter J, Sheidy J, McLin R, Flowers J, Majmudar M, Elgin E, Vilarino V, Lumelsky D, Bhardwaj V, Padula W, Allen JK, Martin SS. Corrie Health Digital Platform for Self-Management in Secondary Prevention After Acute Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005509. doi: 10.1161/CIRCOUTCOMES.119.005509. PMID 31043065
- [Background] Shah LM, Yang WE, Demo RC, Lee MA, Weng D, Shan R, Wongvibulsin S, Spaulding EM, Marvel FA, Martin SS. Technical Guidance for Clinicians Interested in Partnering With Engineers in Mobile Health Development and Evaluation. JMIR Mhealth Uhealth. 2019 May 15;7(5):e14124. doi: 10.2196/14124. PMID 31094337
- [Background] Marvel FA, Wang J, Martin SS. Digital Health Innovation: A Toolkit to Navigate From Concept to Clinical Testing. JMIR Cardio. 2018 Jan 18;2(1):e2. doi: 10.2196/cardio.7586. PMID 31758761
- [Result] Shah LM, Ding J, Spaulding EM, Yang WE, Lee MA, Demo R, Marvel FA, Martin SS. Sociodemographic Characteristics Predicting Digital Health Intervention Use After Acute Myocardial Infarction. J Cardiovasc Transl Res. 2021 Oct;14(5):951-961. doi: 10.1007/s12265-021-10098-9. Epub 2021 May 17. PMID 33999374
- [Result] Shan R, Ding J, Weng D, Spaulding EM, Wongvibulsin S, Lee MA, Demo R, Marvel FA, Martin SS. Early blood pressure assessment after acute myocardial infarction: Insights using digital health technology. Am J Prev Cardiol. 2020 Sep;3:100089. doi: 10.1016/j.ajpc.2020.100089. Epub 2020 Sep 17. PMID 32964212
- [Result] Yang WE, Spaulding EM, Lumelsky D, Hung G, Huynh PP, Knowles K, Marvel FA, Vilarino V, Wang J, Shah LM, Xun H, Shan R, Wongvibulsin S, Martin SS. Strategies for the Successful Implementation of a Novel iPhone Loaner System (iShare) in mHealth Interventions: Prospective Study. JMIR Mhealth Uhealth. 2019 Dec 16;7(12):e16391. doi: 10.2196/16391. PMID 31841115
- [Result] Hung G, Yang WE, Marvel FA, Martin SS. Mobile health application platform 'Corrie' personalises and empowers the heart attack recovery patient experience in the hospital and at home for an underserved heart attack survivor. BMJ Case Rep. 2020 Feb 17;13(2):e231801. doi: 10.1136/bcr-2019-231801. PMID 32071124
- [Result] Marvel FA, Spaulding EM, Lee MA, Yang WE, Demo R, Ding J, Wang J, Xun H, Shah LM, Weng D, Carter J, Majmudar M, Elgin E, Sheidy J, McLin R, Flowers J, Vilarino V, Lumelsky DN, Bhardwaj V, Padula WV, Shan R, Huynh PP, Wongvibulsin S, Leung C, Allen JK, Martin SS. Digital Health Intervention in Acute Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2021 Jul;14(7):e007741. doi: 10.1161/CIRCOUTCOMES.121.007741. Epub 2021 Jul 15. PMID 34261332
- [Derived] Bhardwaj V, Spaulding EM, Marvel FA, LaFave S, Yu J, Mota D, Lorigiano TJ, Huynh PP, Shan R, Yesantharao PS, Lee MA, Yang WE, Demo R, Ding J, Wang J, Xun H, Shah L, Weng D, Wongvibulsin S, Carter J, Sheidy J, McLin R, Flowers J, Majmudar M, Elgin E, Vilarino V, Lumelsky D, Leung C, Allen JK, Martin SS, Padula WV. Cost-effectiveness of a Digital Health Intervention for Acute Myocardial Infarction Recovery. Med Care. 2021 Nov 1;59(11):1023-1030. doi: 10.1097/MLR.0000000000001636. PMID 34534188
- See also: Corrie Health Digital Platform for Self-Management in Secondary Prevention After Acute Myocardial Infarction — http://www.ahajournals.org/doi/full/10.1161/CIRCOUTCOMES.119.005509
- See also: Technical Guidance for Clinicians Interested in Partnering With Engineers in Mobile Health Development and Evaluation — http://mhealth.jmir.org/2019/5/e14124/
- See also: Digital Health Innovation: A Toolkit to Navigate From Concept to Clinical Testing — http://cardio.jmir.org/2018/1/e2
- See also: Sociodemographic Characteristics Predicting Digital Health Intervention Use After Acute Myocardial Infarction — http://link.springer.com/article/10.1007/s12265-021-10098-9
- See also: Strategies for the Successful Implementation of a Novel iPhone Loaner System (iShare) in mHealth Interventions: Prospective Study — http://mhealth.jmir.org/2019/12/e16391
- See also: Mobile health application platform 'Corrie' personalises and empowers the heart attack recovery patient experience in the hospital and at home for an underserved heart attack survivor — http://casereports.bmj.com/content/bmjcr/13/2/e231801.full.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 participants were enrolled in 4 hospitals to receive study intervention. 864 patients' data were pulled from hospital administrative data sets to be the historical comparison group.
Pre-assignment Details: Patients in the historical comparison group were not considered enrolled in this study.
Groups:
- Corrie Digital Health Platform Group: Receives the Corrie Digital Health intervention plus the standard of care
  Corrie Digital Health platform: The Corrie Digital Health platform consists of the Corrie smartphone app for heart attack recovery which is paired with an Apple Watch and Bluetooth-enabled, iHealth blood pressure cuff.
- Historical Comparison Group: Receives the standard of care
Period: Overall Study
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group
Started | 200 | 864
Completed | 200 | 864
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group | Total
Number analyzed (Participants) | 200 | 864 | 1064
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.5) | 65.4 (14.1) | 64.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 336 | 394
  Male | 142 | 528 | 670
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 137 | 561 | 698
  Race: Non-White | 57 | 285 | 342
  Race: Unknown | 6 | 18 | 24
Insurance status [Count of Participants; unit: Participants] — Population: In historical comparison group a primary payer for insurance of "Workers compensation/unknown" considered as "unknown".
  Participants
    Private insurance/PPO/HMO | 110 | 348 | 458
    Medicare | 62 | 428 | 490
    Medicaid | 22 | 45 | 67
    Self-pay | 6 | 11 | 17
    Unknown | 0 | 32 | 32
Marital status [Count of Participants; unit: Participants]
  Married | 117 | 359 | 476
  Not married | 77 | 465 | 542
  Unknown | 6 | 40 | 46
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: 26.6% missing body mass index data for historical control group
  kg/m^2
    number analyzed (Participants) | 200 | 634 | 834
    (all) | 30.6 (5.9) | 29.5 (8.2) | 29.7 (7.9)
Smoking status [Count of Participants; unit: Participants] — Population: 13.2% (114/864) of the participants in the historical comparison group had missing data for smoking status.
  Participants
    number analyzed (Participants) | 200 | 750 | 950
    Current smoker | 57 | 193 | 250
    Former smoker | 53 | 284 | 337
    Never smoker | 90 | 273 | 363
Total Elixhauser comorbidity count [Median (Inter-Quartile Range); unit: Number of comorbidities per patient] — Population: Unweighted, Agency for Healthcare Research and Quality Elixhauser comorbidity count includes 29 comorbidities with no imputation for missing values. 2.5% missing data for the Corrie intervention group and 1.9% missing data for the historical comparison group.
  Number of comorbidities per patient
    number analyzed (Participants) | 195 | 848 | 1043
    (all) | 3 [2 to 5] | 4 [2 to 6] | 4 [2 to 5]
Hospital of Admission [Count of Participants; unit: Participants]
  Johns Hopkins Hospital | 104 | 437 | 541
  Johns Hopkins Bayview Medical Center | 70 | 297 | 367
  Massachusetts General Hospital | 14 | 70 | 84
  Reading Hospital | 12 | 60 | 72
Type of Acute Myocardial Infarction [Count of Participants; unit: Participants]
  NSTEMI | 121 | 676 | 797
  STEMI | 79 | 188 | 267
Intervention (during index admission) [Count of Participants; unit: Participants]
  Percutaneous coronary intervention alone | 131 | 320 | 451
  Coronary artery bypass grafting surgery alone | 44 | 134 | 178
  Both | 8 | 4 | 12
  Neither | 17 | 406 | 423
Length of stay [Median (Inter-Quartile Range); unit: days] | 5 [3 to 10] | 4 [2 to 9] | 4 [3 to 9]
Discharge disposition [Count of Participants; unit: Participants]
  Home | 167 | 555 | 722
  Home care | 18 | 182 | 200
  Skilled nursing facility | 1 | 44 | 45
  Rehabilitation | 12 | 22 | 34
  Hospice/other hospital | 2 | 46 | 48
  AMA/shelters/police custody/unknown | 0 | 15 | 15
Duration of education [Mean (Standard Deviation); unit: years] — Population: 31% missing data for formal education in the Corrie group. This data is not available in the electronic medical record so it could not be obtained for the historical comparison group.
  years
    number analyzed (Participants) | 138 | 0 | 138
    (all) | 14.6 (3.6) |  | 14.6 (3.6)
Household income per year [Median (Inter-Quartile Range); unit: US dollars] — Population: 54.5% missing data on household income for the Corrie intervention group. This data is not available in the electronic medical record so it could not be obtained for the historical comparison group.
  US dollars
    number analyzed (Participants) | 91 | 0 | 91
    (all) | 70,000 [40,000 to 113,000] |  | 70,000 [40,000 to 113,000]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Readmitted Within 30-days Post Hospital Discharge
Description: Number of participants readmitted within 30-days post hospital discharge in the Corrie Digital Health Group as compared to the Historical Standard of Care Comparison group, collected from hospital administrative databases.
Time Frame: 30-days post hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group
Number analyzed (Participants) | 200 | 864
Participants | 13 | 145
Statistical Analysis 1: Comparison: Corrie Digital Health Platform Group vs Historical Comparison Group; Test type: Other; p = 0.018, Regression, Cox — The a priori threshold for statistical significance was <0.05; Adjusting for hospital site and a propensity score inclusive of individual level baseline characteristics; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.26 to 0.88]

2. Secondary Outcome: Cost-effectiveness as Assessed by a Markov Model of Cost-effectiveness
Description: We estimated typical costs associated with readmissions or death of acute myocardial infarction (AMI) patients discharged with standard practices using 2014 US hospital costs from the Agency for Healthcare Research and Quality (AHRQ). The hospital cost (in US dollars) for unplanned 30-day readmission is presented for the Corrie Digital Health Platform Group and the Historical Comparison Group. The reported number is the estimated cost per readmission per participant since the exact cost of the readmission for each patient who was readmitted within 30-days wasn't available. No measure of central tendency is available.
Time Frame: 30 days post hospital discharge
Population: 200 patients enrolled in the Corrie group as compared to data from the historical comparison group as well as model estimates obtained from the literature for the standard of care comparison. Model estimates from the literature were used to supplement information when data was not available from the historical comparison group. The addition of the model estimates from the literature ensured the testing of representative, real-world values.
Measure: Number; unit: US dollars
Groups:
- Corrie Digital Health Platform Group: Receives the Corrie Digital Health intervention plus the standard of care Corrie Digital Health platform: The Corrie Digital Health platform consists of the Corrie smartphone app for heart attack recovery which is paired with an Apple Watch and Bluetooth-enabled, iHealth blood pressure cuff. obtained from the literature.
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group
Number analyzed (Participants) | 200 | 864
US dollars | 17,195 | 27,940
Statistical Analysis 1: Comparison: Corrie Digital Health Platform Group vs Historical Comparison Group; Test type: Other — A Markov Model of cost-effectiveness, based on 30-day readmission rates, was built to assess the Incremental Cost-Effectiveness Ratio (ICER) of adopting the Corrie Platform compared to standard of care for post AMI patients; taking into account the estimated cost of Corrie ($2,750 per patient for a 1-year use term). The reported value is a ratio of the relative cost of intervention compared to the standard of care divided by the change in the outcome, quality-adjusted life years (QALYs); Incremental Cost-Effectiveness Ratio = -7,319 — A negative ICER means the intervention cost is lower than the cost of standard of care, while the denominator was positive. A positive ICER means the intervention cost is greater than the cost of standard of care, while the denominator was positive

3. Secondary Outcome: In-hospital Care Satisfaction as Assessed by a Subset of the Hospital Consumer Assessment of Healthcare Providers and Systems Survey (9 Items)
Description: Among participants in the Corrie Digital Health group, a nine-item five-point Likert scale for assessing in-hospital care satisfaction 3 days post-discharge is used with scoring from 1 "strongly disagree" to 5 "strongly agree", with higher scores meaning participants were more satisfied with the care received. A total score of these nine items is calculated with possible total scores ranging from 9 to 45.
Time Frame: 3 days post hospital discharge
Population: 89 participants completed all the items on the survey, except for one where one person did not fill out the item/question, resulting in 88 being analyzed for that item.
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 89
Participants
  I would recommend this hospital to my friends and family.: Strongly Disagree | 0
  I would recommend this hospital to my friends and family.: Disagree | 0
  I would recommend this hospital to my friends and family.: Neither Disagree nor Agree | 3
  I would recommend this hospital to my friends and family.: Agree | 21
  I would recommend this hospital to my friends and family.: Strongly Agree | 65
  During this hospital stay, the nurses treated me with courtesy and respect.: number analyzed (Participants) | 88
  During this hospital stay, the nurses treated me with courtesy and respect.: Strongly Disagree | 0
  During this hospital stay, the nurses treated me with courtesy and respect.: Disagree | 0
  During this hospital stay, the nurses treated me with courtesy and respect.: Neither Disagree nor Agree | 1
  During this hospital stay, the nurses treated me with courtesy and respect.: Agree | 15
  During this hospital stay, the nurses treated me with courtesy and respect.: Strongly Agree | 72
  During this hospital stay, the nurses listened carefully to me.: Strongly Disagree | 0
  During this hospital stay, the nurses listened carefully to me.: Disagree | 0
  During this hospital stay, the nurses listened carefully to me.: Neither Disagree nor Agree | 2
  During this hospital stay, the nurses listened carefully to me.: Agree | 21
  During this hospital stay, the nurses listened carefully to me.: Strongly Agree | 66
  During this hospital stay, the nurses explained things in a way I could understand.: Strongly Disagree | 0
  During this hospital stay, the nurses explained things in a way I could understand.: Disagree | 0
  During this hospital stay, the nurses explained things in a way I could understand.: Neither Disagree nor Agree | 1
  During this hospital stay, the nurses explained things in a way I could understand.: Agree | 19
  During this hospital stay, the nurses explained things in a way I could understand.: Strongly Agree | 69
  During this hospital stay, the doctors treated me with courtesy and respect.: Strongly Disagree | 0
  During this hospital stay, the doctors treated me with courtesy and respect.: Disagree | 0
  During this hospital stay, the doctors treated me with courtesy and respect.: Neither Disagree nor Agree | 1
  During this hospital stay, the doctors treated me with courtesy and respect.: Agree | 17
  During this hospital stay, the doctors treated me with courtesy and respect.: Strongly Agree | 71
  During this hospital stay, the doctors listened carefully to me.: Strongly Disagree | 0
  During this hospital stay, the doctors listened carefully to me.: Disagree | 1
  During this hospital stay, the doctors listened carefully to me.: Neither Disagree nor Agree | 2
  During this hospital stay, the doctors listened carefully to me.: Agree | 20
  During this hospital stay, the doctors listened carefully to me.: Strongly Agree | 66
  During this hospital stay, the doctors explained things in a way I could understand.: Strongly Disagree | 0
  During this hospital stay, the doctors explained things in a way I could understand.: Disagree | 1
  During this hospital stay, the doctors explained things in a way I could understand.: Neither Disagree nor Agree | 2
  During this hospital stay, the doctors explained things in a way I could understand.: Agree | 21
  During this hospital stay, the doctors explained things in a way I could understand.: Strongly Agree | 65
  The hospital staff talked with me about whether I would have the help I needed after leaving.: Strongly Disagree | 0
  The hospital staff talked with me about whether I would have the help I needed after leaving.: Disagree | 1
  The hospital staff talked with me about whether I would have the help I needed after leaving.: Neither Disagree nor Agree | 3
  The hospital staff talked with me about whether I would have the help I needed after leaving.: Agree | 33
  The hospital staff talked with me about whether I would have the help I needed after leaving.: Strongly Agree | 52
  Before giving any new medications, hospital staff described clearly potential side effects.: Strongly Disagree | 0
  Before giving any new medications, hospital staff described clearly potential side effects.: Disagree | 9
  Before giving any new medications, hospital staff described clearly potential side effects.: Neither Disagree nor Agree | 14
  Before giving any new medications, hospital staff described clearly potential side effects.: Agree | 28
  Before giving any new medications, hospital staff described clearly potential side effects.: Strongly Agree | 38

4. Secondary Outcome: In-hospital Care Satisfaction as Assessed by a Subset of the Hospital Consumer Assessment of Healthcare Providers and Systems Survey (Summary Score)
Description: as for outcome 3
Time Frame: 3 days post hospital discharge
Population: 89 participants completed the items on the survey.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 89
score on a scale | 43 [40 to 45]

5. Secondary Outcome: In-hospital Care Satisfaction as Assessed by a Subset of the Hospital Consumer Assessment of Healthcare Providers and Systems Survey (1 Dichotomous Item)
Description: Among participants in the Corrie Digital Health group, one additional item, not on the five-point Likert scale, for assessing in-hospital care satisfaction 3 days post-discharge asked if they received information in writing about what symptoms or health problems to look out for after leaving the hospital (Yes/No).
Time Frame: 3 days post hospital discharge
Population: 88 participants completed this item on the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 88
Participants
  Yes | 79
  No | 9

6. Secondary Outcome: In-hospital Care Satisfaction as Assessed by a Subset of the Hospital Consumer Assessment of Healthcare Providers and Systems Survey (1 Continuous Item)
Description: Among participants in the Corrie Digital Health group, one additional item, not on the five-point Likert scale, for assessing in-hospital care satisfaction 3 days post-discharge asked them to provide an overall hospital rating on a 1-10 sliding scale with a higher score indicating a higher overall hospital rating.
Time Frame: 3 days post hospital discharge
Population: 68 participants completed this item on the survey.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 68
score on a scale | 10 [9 to 10]

7. Secondary Outcome: Perceived Usability of Corrie as Assessed by the Systems Usability Scale
Description: Among participants in the Corrie Digital Health group, a 10-item five-point Likert scale for assessing systems usability of Corrie both 3 and 30 days post-discharge is used with scoring from 0 to 4 and higher scores meaning patients perceive the system as having global usability. The total score reference range is from 0 to 100, where lower scores indicate lower perceived application usability.
Time Frame: 3 and 30 days post hospital discharge
Population: At 3 days post discharge, 87 participants completed the survey, while at 30 days post-discharge 104 participants completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 104
score on a scale
  3 days post-discharge: number analyzed (Participants) | 87
  3 days post-discharge | 58.6 (11.5)
  30 days post-discharge | 57.6 (11.6)

8. Secondary Outcome: Perceived Corrie App Satisfaction as Assessed by a Study Team Developed Scale
Description: Among participants in the Corrie Digital Health group, a five-item five-point Likert scale for assessing participant satisfaction with Corrie as a tool to improve acute myocardial infarction recovery 3 and 30 days post-discharge is used with scoring from 1 to 5 and higher scores meaning more satisfaction with Corrie. Total possible scores ranging from 5 to 25, where higher scores indicate greater Corrie app satisfaction.
Time Frame: 3 and 30 days post hospital discharge
Population: 80 participants completed the survey at 3 days post-discharge and 99 completed the survey at 30 days post-discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 99
score on a scale
  3 days post-discharge: number analyzed (Participants) | 80
  3 days post-discharge | 18.29 (3.75)
  30 days post-discharge | 17.65 (3.68)

9. Secondary Outcome: User Engagement With Corrie App as Assessed by the User Engagement Scale
Description: Among participants in the Corrie Digital Health group, a 29-item five-point Likert scale for assessing the subjective experience of user engagement with Corrie 30 days post discharge is used with scoring ranging from 1 to 5 and higher scores reflecting higher perceived user engagement. The total subjective user engagement score was calculated by diving the sum of all items by 29, resulting in a range of potential total scores from 1 to 5.
Time Frame: 30 days post hospital discharge
Population: 102 participants completed the survey at 30 days post-discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 102
score on a scale | 3.36 (0.57)

10. Secondary Outcome: User Engagement With Corrie Health App as Assessed by the Total Number of Interactions Per Participant in the Smartphone App, Collected Via Corrie Health Platform User Analytics
Description: The total number of app interactions is a behavioral manifestation of user engagement and is monitored through app usage data. The total number of app interactions consisted of: number of BP, heart rate,weight, mood, and step count recordings; number of medications tracked; and number of educational articles and videos viewed over the study period.
Time Frame: Throughout the study period for app usage up to 30 days post-discharge from the hospital
Population: Following deployment of Corrie backend capabilities (the Corrie backend was not set up to capture application interactions for the first 34 participants enrolled), 83% (138/166) of Corrie users had captured application interactions (i.e. used the Corrie platform at least once over the 30-day study and subsequently connected to WiFi or cellular data to connect with the backend).
Measure: Median (Inter-Quartile Range); unit: Number of app interactions/participant
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 138
Number of app interactions/participant | 213 [35 to 428]

11. Secondary Outcome: User Engagement With Corrie Health App as Assessed by the Overall Amount of Time Spent Using the App, Collected Via Corrie Health Platform App User Analytics
Description: The overall amount of time (days) spent using the app is a behavioral manifestation of user engagement and is monitored through app usage data and collected via Corrie Health Platform app user analytics.
Time Frame: Throughout the study period for app usage up to 30 days post-discharge from the hospital
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 138
days | 12 [2 to 29]

12. Secondary Outcome: Patient Activation as Assessed by the Patient Activation Measure
Description: Among participants in the Corrie Digital Health group, the 10-item five-point Likert scale for assessing patient activation 3 and 30 days post-discharge is used with scoring ranging from 1 to 5 and higher scores indicating the patient possesses the necessary knowledge, skills, and confidence needed for self-care. The total score reference range is from 0 to 100, where lower scores indicate lower patient activation.
Time Frame: 3 and 30 days post hospital discharge
Population: At 3-days post discharge only 94 participants completed the survey while at 30 days post-discharge 103 participants completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 103
score on a scale
  3 days post-discharge: number analyzed (Participants) | 94
  3 days post-discharge | 71.9 (15.7)
  30 days post-discharge | 71.7 (16.6)

13. Secondary Outcome: Cardiac Medication Adherence as Assessed by the Adherence to Refills and Medications Scale Subscale
Description: Among participants in the Corrie Digital Health group, the eight-item four-point Likert scale for assessing cardiac medication adherence 30 days post-discharge is used with scoring ranging from 1 to 4 and lower scores indicating better adherence. Total possible scores could range from 8 to 32 with lower scores indicating better adherence. The total cardiac medication adherence score was dichotomized into completely cardiac medication adherent and near completely cardiac medication adherent, based on the median score.
Time Frame: 30 days post hospital discharge
Population: 102 participants completed the survey at 30 days post-discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 102
Participants
  Complete Adherence | 81
  Near Complete Adherence | 21

14. Secondary Outcome: Cardiac Medication Adherence as Assessed by Smartphone App Usage Data
Description: Cardiac medication adherence (beta-blockers, anti-platelets, statins) is measured from the smartphone app usage data as the percentage of cardiac medications marked as "taken".
Time Frame: Throughout the study period for app usage up to 30 days post-discharge from the hospital
Population: 135 patients who had app interaction data specific to cardiovascular disease (CVD) medications (beta-blocker, anti-platelet, statin) from admission through 30 days post-discharge.
Measure: Number (95% Confidence Interval); unit: percentage of any CVD meds marked taken
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 135
percentage of any CVD meds marked taken | 87 [82 to 92]

15. Secondary Outcome: Medication Adherence as Assessed by Smartwatch App Usage Data
Description: Medication adherence is measured from the smartwatch app usage data as percent of pills marked as taken.
Time Frame: Throughout the study period for app usage up to 30 days post-discharge from the hospital
Population: Unable to differentiate smartwatch app usage data from smartphone app usage data. Thus, results assessing medication adherence by smartwatch app is provided under as "assessed by smartphone app usage data" (Outcome 13).
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants Who Had Emergency Department Visits Within 30-days Post Hospital Discharge
Description: Number of participants who had Emergency department visits (at Johns Hopkins Hospital and Johns Hopkins Bayview Medical Center) within 30-days post hospital discharge, that did not result in readmission, in the Corrie Digital Health Group as compared to the Historical Standard of Care Comparison group, collected from hospital administrative databases.
Time Frame: 30 days post hospital discharge
Population: 908 patients were enrolled at Johns Hopkins Hospital and Johns Hopkins Bayview Medical Center across both the Corrie intervention group (n=174) and historical comparison group (n=734). 80 of the patients had an emergency department visit within 30-days of discharge that resulted in a readmission and were excluded from this analysis. Hence, a total of 828 participants were included in the analysis across the Corrie intervention group (n=164) and the historical comparison group (n=664).
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group
Number analyzed (Participants) | 164 | 664
Participants | 13 | 39
Statistical Analysis 1: Comparison: Corrie Digital Health Platform Group vs Historical Comparison Group; Test type: Other; p = 0.33, Regression, Cox — The a priori threshold for statistical significance was <0.05; Adjusting for hospital site and a propensity score inclusive of individual level baseline characteristics; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.69 to 2.98]

17. Secondary Outcome: Number of Hospital Observations
Description: Number of hospital observations within 30-days post hospital discharge in the Corrie Digital Health Group as compared to the Historical Standard of Care Comparison group, collected from hospital administrative databases.
Time Frame: 30 days post hospital discharge
Population: Unable to obtain this data from hospital administrative data sets. Data was not collected.
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Attendance of Follow-up Appointments as Assessed by Post-discharge Survey Developed by Study Team
Description: Among participants in the Corrie Digital Health group, the investigators are querying participants in the surveys sent out 30 days post-discharge as to whether participants attended an appointment with a primary care provider, cardiologist, and/or cardiac rehab. A point is given to each appointment attended with scores raging from 0 to 3.
Time Frame: 30 days post hospital discharge
Population: 104 participants completed this survey question at 30 days post-discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 104
Participants
  3 appointments attended | 34
  2 appointments attended | 48
  1 appointment attended | 19
  0 appointments attended | 3

19. Secondary Outcome: Number of Readmitted Participants Who Had Recurrent Myocardial Infarctions
Description: Number of readmitted participants who had Recurrent myocardial infarctions in the Corrie Digital Health Group. Participants who had an all-cause 30-day readmission in the Corrie group, as identified by hospital administrative datasets, underwent further chart review to determine if the cause of readmission was a recurrent myocardial infarction.
Time Frame: 30 days post hospital discharge
Population: Total of 13 participants in the Corrie group who were readmitted within 30 days of discharge. Unable to obtain reason for readmission from the hospital administrative data sets. Thus, data on whether 30-day readmissions were due to recurrent myocardial infarction were not available for the historical comparison group. Chart review, to obtain this reason for readmission as done with the Corrie group, was not possible for the historical comparison group.
Measure: Count of Participants; unit: Participants
Arm/Group | Corrie Digital Health Platform Group
Number analyzed (Participants) | 13
Participants | 0

20. Secondary Outcome: Number of Deaths Within 30 Days Post Hospital Discharge
Description: Death within 30-days post hospital discharge in the Corrie Digital Health Group as compared to the Historical Standard of Care Comparison group, collected from hospital administrative databases.
Time Frame: 30 days post hospital discharge
Population: Unable to obtain data from hospital administrative data sets. Data was not collected.
Arm/Group | Corrie Digital Health Platform Group | Historical Comparison Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment in the hospital to 30 days post-discharge, for the Corrie Digital Health Platform group.
Description: While 30-day hospital readmission data was collected for both the Corrie Digital Health Platform and Historical Comparison groups this data is not listed here for the Historical Comparison group because they were not enrolled participants. All-cause mortality data could not be obtained from hospital administrative databases. It was reported to the study team by the participant's family member. This explains why outcome measure 20 has no data but 1 mortality reported here.
Groups:
- Corrie Digital Health Platform Group: Receives the Corrie Digital Health intervention plus the standard of care
  Corrie Digital Health platform: The Corrie Digital Health platform consists of the Corrie smartphone app for heart attack recovery which is paired with an Apple Watch and Bluetooth-enabled, iHealth blood pressure cuff.
  The sample size for reporting of adverse events is 216. 200 Corrie patients that finished the study plus 16 who were consented but later withdrew or were withdrawn from the study.
Arm/Group | Corrie Digital Health Platform Group
All-Cause Mortality (participants affected / at risk) | 1/200
Serious Adverse Events (participants affected / at risk) | 13/200
Other Adverse Events (participants affected / at risk) | 1/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Corrie Digital Health Platform Group (N=200)
Inpatient hospital readmission within 30 days post-discharge (General disorders) | 13 — Number of participants that were readmitted within 30 days post-discharge among the 200 Corrie participants that completed the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Corrie Digital Health Platform Group (N=200)
Bruising (General disorders) | 1 — Report of bruising on participant forearm, where the Apple Watch was located. Bruising was reported in other locations. The participant was on blood thinners, with a history of bruising. It is uncertain if the Apple Watch contributed to bruising.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03760796/Prot_SAP_001.pdf
  • Informed Consent Form (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT03760796/ICF_000.pdf